CLINICAL TRIAL: NCT05716126
Title: Study Evaluating the Mass Balance and Biotransformation of Single Dose [14C]Iruplinalkib (WX-0593) In Healthy Male Volunteers
Brief Title: Single Dose Mass Balance Study With [14C]Iruplinalkib (WX-0593) In Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WX0593-005
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14]Iruplinalkib(WX-0593) 120 mg(orla solution) (Experimental): Volunteer will receive a single oral dose of 120 mg [14C]Iruplinalkib (WX-0593) administered by mouth, as a solution.
  Interventions: Drug: [14C]Iruplinalkib (WX-0593)

INTERVENTIONS:
Drug: [14C]Iruplinalkib (WX-0593) — Volunteer will receive a single oral dose of 120 mg [14C]Iruplinalkib (WX-0593) as a solution on Day 1

SUMMARY:
This is an open-label, single dose, mass balance and biotransformation study conducted at 1 study center in China. This study will evaluate the absorption, distribution, metabolism, and elimination (ADME), mass balance, safety, and tolerability of a single dose of intravenously administered [14C]Iruplinalkib (WX-0593) in Chinese healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old (inclusive) healthy male volunteers;
* Body mass index 19.0-26.0 kg/m 2 (inclusive) and body weight ≥50 kg;
* The volunteer has fully given informed consent to the study and voluntarily signed the informed consent form prior to trial.

Exclusion Criteria:

* Physical examination, vital signs, laboratory tests (routine blood test, urinalysis, stool + occult blood test, blood biochemistry, blood coagulation, and thyroid function), ophthalmic examination (slit lamp exam, intraocular pressure, and fundus imaging), 12-lead electrocardiogram, chest X-ray (posteroanterior view), and abdominal ultrasound results that are determined abnormal and clinically significant by the investigator during screening;
* Positive for HBsAg, HBeAg, HCV antibody, HIV antibody, or syphilis antibody;
* Has taken any prescribed medication and herbal medicine within 1 month prior to dosing, or has taken over-the-counter medications or food supplements (e.g. Vitamins or calcium) within 2 months prior to dosing;
* Has participated in clinical trials of any other drug within 3 months prior to dosing;
* Previous heart disease or family history of heart disease, such as organic heart disease, heart failure, myocardial infarction, angina, irreducible arrhythmia, torsades de pointes, ventricular tachycardia, or long QT syndrome;
* Major surgery within 6 months prior to dosing or surgical incision is not completely healed; Major surgery includes but is not limited to surgery with any significant risk of bleeding, prolonged general anesthesia, biopsy or significant traumatic injury;
* Any history of severe clinical illness or disease and conditions that are judged by the investigator to potentially affect the results of the study or disease and history of disease that can reduce treatment adherence (including but not limited to cardiovascular, liver, kidney, gastrointestinal, immune, urinary, blood, endocrine, metabolic, mental, and neurological diseases as well as cancer), especially a history of dysphagia, gastrointestinal ulcers or any gastrointestinal disorders that affect drug absorption;
* Known allergy to two or more substances; Or potential allergy to the test drug or its excipients in the judgment of the investigator, or allergy to any food ingredients, or special requirements for diet and inability to consume a uniform diet;
* Hemorrhoids or perianal disease with regular/current bleeding;
* Habitual constipation, diarrhea, irritable bowel syndrome, or inflammatory bowel disease;
* Consumed over 14 units of alcohol (1 unit = 360 mL beer or 45 mL of liquor with 40% alcohol or 150 mL wine) weekly within 6 months prior to screening or breath alcohol test result of ≥20 mg/dL;
* Consumed more than 5 cigarettes daily within 3 months prior to screening or inability to quit smoking during the study;
* Consumed soft drugs (e.g. Marijuana, MDMA, ketamine or magu/yaba) within 3 months prior to dosing or hard drugs (E.g. Cocaine, heroin, or methamphetamine) within 1 year prior to dosing or positive for urine drug test;
* Habitually consumed grapefruit or grapefruit juice, or excessively consumed tea, coffee, alcohol and/or drinks containing caffeine or alcohol and unable to quit during hospitalization, or frequent strenuous exercise and other factors that affect drug absorption, distribution, metabolism, and excretion;
* Consumed any food or drink rich in xanthine (e.g. Animal organs, chocolate, tea, coffee or coke) within 48 hr prior to dosing, or any grapefruit or products containing grapefruit within 48 hr prior to dosing;
* Donated blood within 3 months prior to dosing or lost >400 mL of blood or received blood transfusion within 8 weeks prior to dosing;
* Plan to conceive during and within 1 year after trial completion, or disagree with taking strict contraceptive measures (by the volunteer and his spouse) during and within 1 year after trial completion;
* Work in conditions with long-term radiation exposure, or had significant radiation exposure (received ≥2 chest/abdominal CT, or ≥3 other x-ray exams) within 1 year of signing the informed consent, or participated in radioactive drug trials, or plan to have radiation exposure within 1 year after trial completion.
* Any other factors which in the judgment of the investigator render the volunteer unsuitable for the trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Metabolic profiling for iruplinalkib(WX-0593) will be determined in plasma samples. | Assessments will be made up to 3 days post dose.
  Percent (%) of each radiolabeled drug-related material (parent and each metabolite) will be determined in plasma, urine and feces.
Metabolic profiling for iruplinalkib(WX-0593) will be determined in urine samples. | Assessments will be made up to 3 days post dose.
  Percent (%) of each radiolabeled drug-related material (parent and each metabolite) will be determined in urine.
metabolic profiling for iruplinalkib(WX-0593) will be determined in fecal samples. | Assessments will be made up to 3 days post dose.
  Percent (%) of each radiolabeled drug-related material (parent and each metabolite) will be determined in feces.
Total Radioactivity in Feces | Assessments will be made up to 14 days post dose.
  Cumulative amount was calculated as sum of feces drug concentration in sample volume for each collection interval.
Total Radioactivity in Urine | Assessments will be made up to 14 days post dose.
  Cumulative amount was calculated as sum of urine drug concentration in sample volume for each collection interval.

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Assessments will be made up to 28 days post dose.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China